CLINICAL TRIAL: NCT05898685
Title: Effect of a Single Session of Intermittent Hypoxia on Hematological Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Sophie Lalande, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-09-0015
Record Dates: First submitted 2023-05-29; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Intermittent Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent hypoxia (Experimental): The intermittent hypoxia protocol will consist of eight 4-minute hypoxic cycles (arterial oxygen saturation of 80%) interspersed with normoxic cycles to resaturation.
  Interventions: Behavioral: Intermittent hypoxia
- Intermittent normoxia (Sham Comparator): The intermittent normoxia protocol will consist of eight 4-minute normoxic cycles (compressed air) interspersed with 1-minute normoxic cycles (room air).
  Interventions: Behavioral: Intermittent normoxia

INTERVENTIONS:
Behavioral: Intermittent hypoxia — The intermittent hypoxia protocol will consist of eight 4-minute hypoxic cycles (arterial oxygen saturation of 80%) interspersed with normoxic cycles to resaturation.
  Arms: Intermittent hypoxia
Behavioral: Intermittent normoxia — The intermittent normoxia protocol will consist of eight 4-minute normoxic cycles (compressed air) interspersed with 1-minute normoxic cycles (room air)
  Arms: Intermittent normoxia

SUMMARY:
The purpose of the study is to determine the effect of a single exposure of intermittent hypoxia on erythropoietin levels and hemoglobin mass in young adults, older adults and patients with type 2 diabetes.

DETAILED DESCRIPTION:
Cardiorespiratory fitness, assessed by measuring maximal oxygen consumption (VO2max), has a potential to predict cardiovascular disease and mortality risk to a greater extent than smoking, hypertension, type 2 diabetes or high cholesterol levels. Oxygen transport from the lungs to the exercising muscles is achieved through the binding of oxygen to hemoglobin, an iron-containing protein in the red blood cell. Therefore, hemoglobin mass represents the oxygen-carrying capacity of the blood and strongly correlates with VO2max. Patients with type 2 diabetes have serious impairments in cardiorespiratory fitness, as observed through a 20% lower VO2max than individuals matched for age, weight and physical activity levels. The investigators previously showed that a lower hemoglobin mass limits oxygen-carrying capacity and contributes to the lower VO2max in patients with type 2 diabetes. Thus, interventions that can increase hemoglobin mass should result in improved oxygen-carrying capacity and VO2max in patients with type 2 diabetes. While the majority of patients with type 2 diabetes are aware of their need to perform exercise to improve their VO2max, less than 1/3 of patients meet recommended levels of physical activity. There is therefore an urgent need to develop alternative interventions that improve VO2max, as even minimal improvements in VO2max significantly decrease mortality risk in unfit individuals.

Hypoxia deprives the body of adequate oxygen supply at the tissue level which stimulates the release of erythropoietin (EPO), the peptide hormone regulating red blood cell production, in order to restore oxygen supply to the tissues. Following a rise in EPO levels, it takes 5-6 days for a newly created reticulocyte to mature into a red blood cell, and to observe an increased hemoglobin mass. Increases in EPO levels have been observed to reach maximum values approximately 2-3 h after continuous hypoxic exposure lasting between 90 minutes and 3 hours. It has consequently been suggested that intermittent hypoxia, consisting of alternating few minutes of breathing hypoxic air with few minutes of breathing normoxic air, would provide a stimulus sufficient to stimulate an increase in EPO levels and hematological variables. Only one study measured both EPO levels and hematological changes in responses to intermittent hypoxia. Elite distance runners completed 4 weeks of intermittent hypoxia consisting of 5:5-minutes hypoxia-to-normoxia ratio for 70 min, 5 times/week. The fraction of inspired oxygen gradually declined from 0.12 to 0.10%. The authors did not observe any increase in EPO levels or hemoglobin concentration. However, there were several methodological limitations that could explain these findings. First, hemoglobin concentration is dependent on plasma volume and is therefore greatly influenced by hydration status, and correlates only to a modest extent with red blood cell mass. On the other hand, hemoglobin mass is reported in grams and is a more direct measure of oxygen-carrying capacity. Second, EPO measurements were performed at the same time of day to minimize any circadian variability in EPO levels, which likely prevented the detection of a rise in EPO within the first few hours following the exposure to intermittent hypoxia. Therefore, the purpose of the present study is to determine the effect of a single exposure of intermittent hypoxia on EPO levels and hemoglobin mass in healthy individuals. The cardiovascular and ventilatory responses to a single exposure of intermittent hypoxia will also be determined. If intermittent hypoxia improves oxygen-carrying capacity, the next step will be to apply this intervention to patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years old
* Adults with type 2 diabetes aged 30 to 80 years old

Exclusion Criteria:

* Have high blood pressure (above 140/90 mmHg)
* Are smokers
* Are pregnant
* Have a history of cardiovascular disease, diabetes or lung disease
* Are taking more than one antihypertensive medication
* Are taking insulin or more than one antihypertensive medication
* Have poorly controlled diabetes: HbA1c levels ˃ 9%
* Have been previously diagnosed with diabetic complications (nephropathy, neuropathy, retinopathy) by their family doctor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in erythropoietin levels | Measured before and 4.5 hours after intermittent hypoxia
  Hormone that regulates red blood cell production

CONTACTS AND LOCATIONS:
Locations (1):
- The Unviersity of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wojan F, Stray-Gundersen S, Zhao J, Lalande S. Impaired erythropoietin response to hypoxia in type 2 diabetes. Acta Diabetol. 2024 Jul;61(7):925-932. doi: 10.1007/s00592-024-02269-2. Epub 2024 Apr 4. PMID 38570345